CLINICAL TRIAL: NCT06330766
Title: Impact of Targeted Preoperative Dental Screening on Post-procedural Risk of Infective Endocarditis in Patients Undergoing Transcatheter Aortic Valve Implantation: a Prospective Observational Study
Brief Title: Impact of Preoperative Dental Screening in Reducing Infective Endocarditis Risk in Transcatheter Aortic Valve Implantation Patients
Acronym: DENTAVI
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jordi Dahl, Associate Professor, Chief physician in charge of cardiology imaging, Odense University Hospital
Other Study IDs: PET24
Record Dates: First submitted 2024-02-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Transcatheter Aortic Valve Implantation; Dental; Endocarditis
Keywords: Transcatheter aortic valve implantation; TAVI; Preoperative dental screening; Infectious endocarditis
MeSH Terms: conditions — Endocarditis; Endocarditis, Subacute Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No preoperative dental screening: No preoperative dental screening in patients undergoing TAVI
  Interventions: Procedure: No preoperative dental screening
- Mandatory preoperative dental screening: Mandatory preoperative dental screening in patients undergoing TAVI

INTERVENTIONS:
Procedure: No preoperative dental screening — Discontinuance of mandatory preoperative dental screening prior TAVI which also can include oral surgery.
  Groups: No preoperative dental screening

SUMMARY:
In Odense University Hospital preoperative dental screening (PDS) protocol for patients treated with Transcatheter Aortic Valve Implantation (TAVI) was changed from mandatory to targeted PDS to between June 2023 to october 2023. The investigators will therefore compare the risk of IE before june 2023 and after october 2023.

DETAILED DESCRIPTION:
Infective endocarditis (IE), a condition linked with significant mortality and morbidity rates, is particularly concerning for patients with prosthetic left-sided valves.

These patients face an elevated IE risk, estimated at about 1% annually in tertiary care settings, cumulatively impacting around one in every 20 patients over a decade.

In line with this, both the American Heart Association (AHA) and the European Society of Cardiology (ESC) strongly advocate for the elimination of potential dental sepsis sources at least two weeks before prosthetic valve implantation, except in urgent cases.

These guidelines, while not grounded in randomized trials, largely draw upon registry data detailing IE incidence among surgical aortic valve replacement (SAVR) patients.

In a recent study the investigators found no difference in risk of IE when comparing mandatory preoperative dental screening (MPDS) with no preoperative dental screening (NPDS).

Thus, this prospective registry-based observational before-and-after study aims to investigate the impact of different preoperative dental screening practices on the risk of IE in patients undergoing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAVI

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing TAVI from Oktober 2023 to January 2026 from Odense University Hospital and Aalborg University Hospital compared with same type of patients from the same centers from the period January 2020 to June 2023.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Infectious Endocarditis | Through study completion, an average of 1 year
  Infectious endocarditis diagnosed by healthcare professionals

SECONDARY OUTCOMES:
Number of Participants undergoing Oral surgical procedure at dental screening | Through study completion, an average of 1 year
  Number of oral surgical procedure performed in patients as part of the dental screening
Number of Participants undergoing Tooth extraction at dental screening | Through study completion, an average of 1 year
  Number of Tooth extraction procedure performed in patients as part of the dental screening
The different Bacteria types causing the infectious endocarditis assessed by blood culture | Through study completion, an average of 1 year
  Reporting all the different bacteria type causing infectious endocarditis, including the rate of each bacteria.
Number patients with Bacteremia assessed by positive blood culture | Through study completion, an average of 1 year
  Cases of bacteremia in the population.
Number of Participants with IE caused by bacteria from oral foci | Through study completion, an average of 1 year
  Infectious Endocarditis caused by bacteria from oral foci
Number of Participants with Cardiac implantable electronic device risk of IE | Through study completion, an average of 1 year
  Cardiac implantable electronic device risk of IE

CONTACTS AND LOCATIONS:
Overall Officials: Jordi S Dahl, MD,PhD,DMSc, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Cardiology Department, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from this study, encompassing both individual participant information and a comprehensive data dictionary that defines each field, will be accessible to interested parties. Specifically, we'll be sharing deidentified participant data paired with the mentioned data dictionary. Study protocol and statistical analysis plan will be provided. Prospective researchers can anticipate data availability concurrent with the publication of our findings. To gain access, reach out to Lytfi.Krasniqi@rsyd.dk. Data will be shared with researchers whose proposed use has received approval. Access will be granted primarily for the replication of the results presented in our study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: To be announced
Access Criteria: A signed data access agreement, compliant with regional legislation and data authority requirements, must be obtained prior to data release.

REFERENCES:
- [Background] Que YA, Moreillon P. Infective endocarditis. Nat Rev Cardiol. 2011 Jun;8(6):322-36. doi: 10.1038/nrcardio.2011.43. Epub 2011 Apr 12. PMID 21487430
- [Background] Piper C, Korfer R, Horstkotte D. Prosthetic valve endocarditis. Heart. 2001 May;85(5):590-3. doi: 10.1136/heart.85.5.590. No abstract available. PMID 11303018
- [Background] Ostergaard L, Valeur N, Ihlemann N, Smerup MH, Bundgaard H, Gislason G, Torp-Pedersen C, Bruun NE, Kober L, Fosbol EL. Incidence and factors associated with infective endocarditis in patients undergoing left-sided heart valve replacement. Eur Heart J. 2018 Jul 21;39(28):2668-2675. doi: 10.1093/eurheartj/ehy153. PMID 29584858
- [Background] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Background] Delgado V, Ajmone Marsan N, de Waha S, Bonaros N, Brida M, Burri H, Caselli S, Doenst T, Ederhy S, Erba PA, Foldager D, Fosbol EL, Kovac J, Mestres CA, Miller OI, Miro JM, Pazdernik M, Pizzi MN, Quintana E, Rasmussen TB, Ristic AD, Rodes-Cabau J, Sionis A, Zuhlke LJ, Borger MA; ESC Scientific Document Group. 2023 ESC Guidelines for the management of endocarditis. Eur Heart J. 2023 Oct 14;44(39):3948-4042. doi: 10.1093/eurheartj/ehad193. No abstract available. PMID 37622656
- [Background] Mentias A, Girotra S, Desai MY, Horwitz PA, Rossen JD, Saad M, Panaich S, Kapadia S, Sarrazin MV. Incidence, Predictors, and Outcomes of Endocarditis After Transcatheter Aortic Valve Replacement in the United States. JACC Cardiovasc Interv. 2020 Sep 14;13(17):1973-1982. doi: 10.1016/j.jcin.2020.05.012. PMID 32912457
- [Background] Butt JH, Ihlemann N, De Backer O, Sondergaard L, Havers-Borgersen E, Gislason GH, Torp-Pedersen C, Kober L, Fosbol EL. Long-Term Risk of Infective Endocarditis After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2019 Apr 9;73(13):1646-1655. doi: 10.1016/j.jacc.2018.12.078. PMID 30947917
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e72-e227. doi: 10.1161/CIR.0000000000000923. Epub 2020 Dec 17. No abstract available. PMID 33332150
- [Background] Buckley AJ, Hensey M, O'Connor S, Maree A. Dental screening prior to transcatheter versus surgical aortic valve replacement: International Survey of Current Practices. Catheter Cardiovasc Interv. 2023 Jul;102(1):176-177. doi: 10.1002/ccd.30675. Epub 2023 May 7. No abstract available. PMID 37149755
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Krasniqi L, Schodt Riber LP, Nissen H, Terkelsen CJ, Andersen NH, Freeman P, Povlsen JA, Gerke O, Clavel MA, Dahl JS. Impact of mandatory preoperative dental screening on post-procedural risk of infective endocarditis in patients undergoing transcatheter aortic valve implantation: a nationwide retrospective observational study. Lancet Reg Health Eur. 2023 Nov 22;36:100789. doi: 10.1016/j.lanepe.2023.100789. eCollection 2024 Jan. PMID 38188272